CLINICAL TRIAL: NCT04426500
Title: Use of Perioperative Pain Blocks In Urological Surgery: A Phase III Randomized Single Blind Single Center Three Arm Non-inferiority Trial
Brief Title: Use of Perioperative Pain Blocks In Urological Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Reza Mehrazin, Assistant Professor, Urologic Oncology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GCO 19-1532; NCI-2019-08790 (Registry Identifier: National Cancer Institute)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Results first posted 2022-05-06 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative; Nerve Block; Robotic Surgical Procedures
Keywords: Phase III; Randomized; Single blind; Single Center; Three arm; Non-inferiority
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: This is a single-center, single-blinded, (stratified) randomized placebo-controlled three-arm non-inferiority trial with 2:2:1 allocation ratio.
  People who meet eligibility requirements and provide informed consent will be randomly allocated to 3 groups to receive either UTAP, LTAP or Placebo with a 2:2:1 allocation ratio. The allocation sequence will be stratified by type of surgery (prostatectomy or partial nephrectomy) using stratified block randomization with randomly varying block sizes. Random permuted blocks sizes within stratification groups will be used to minimize the chance of selection bias. Investigators will be blinded to the size of each block with only the study statistician responsible for generating the randomization list knowing this information.
Who Masked: Participant
Masking Description: A randomization service called Sealedenvelope.com available at https://www.sealedenvelope.com/simple-randomiser/v1/ will be used for allocation concealment to ensure that retrieval of the treatment group assignment is only revealed to appropriate team members on a real time basis after each new patient has been screened and consented. This service allows for allocation concealment that would not be possible if the entire randomization list was made available to team members at the beginning of the study. The security and integrity of the codes used by Sealedenvelope.com follows the Food and Drug Administration (FDA) standards for electronic records and follows the International Conference on Harmonisation Good Clinical Practice (ICH GCP) guidelines.
  Participants will be blinded to group allocation throughout the study. Due to the nature of the intervention, it is not possible to blind the investigator to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo/Local Anesthesia (Placebo Comparator): Direct injection of 0.25% bupivacaine into surgical wounds
  Interventions: Drug: Bupivacain
- Ultrasound-guided transversus abdominus plane (UTAP) block (Active Comparator): 30mL of 0.25% bupivacaine will be administered to bilateral TAP using ultrasound guidance in prostatectomies. 40ml 0.25% bupivacaine unilateral will be administered in nephrectomy patients (weight based dosage permitting).
  Interventions: Drug: Bupivacain; Drug: Ultrasound-guided transversus abdominus plane block
- Laparoscopic-guided transversus abdominus plane (LTAP) block (Experimental): 30mL of 0.25% bupivacaine will be administered to bilateral TAP using laparoscopic guidance in prostatectomies. 40ml 0.25% bupivacaine unilateral will be administered in nephrectomy patients (weight based dosage permitting).
  Interventions: Drug: Bupivacain; Drug: Laparoscopic-guided transversus abdominus plane block

INTERVENTIONS:
Drug: Bupivacain — Direct injection of 0.25% bupivacaine into surgical wounds
  Other Names: Local anesthesia
Drug: Ultrasound-guided transversus abdominus plane block — bilateral TAP using ultrasound guidance in prostatectomies
  Other Names: UTAP
  Arms: Ultrasound-guided transversus abdominus plane (UTAP) block
Drug: Laparoscopic-guided transversus abdominus plane block — bilateral TAP using laparoscopic guidance in prostatectomies
  Other Names: LTAP
  Arms: Laparoscopic-guided transversus abdominus plane (LTAP) block

SUMMARY:
The study team aims to prospectively compare Placebo (local administration), ultrasound-guided transversus abdominis plane (UTAP) blocks, and laparoscopic-guided transversus abdominis plane (LTAP) blocks in patients undergoing robotic surgery of the prostate and kidney. The study team expects to be able to equally efficiently administer the blocks using direct visualization and ultrasound guidance. The study team expects that a negative result would obviate the need for longer operative time by eliminating the need for the separate ultrasound guided block while a positive result would demonstrate the increased utility of preoperative ultrasound blocks in managing postoperative pain.

DETAILED DESCRIPTION:
Currently, ultrasound-guided transversus abdominis plane (UTAP) blocks (regional anesthetic blocks) are being employed for the care of urological surgery patients. Local and regional anesthesia is commonly used throughout surgical fields. However, ultrasound-guidance can be challenging, particularly in larger, obese patients. It is unknown how such techniques compare to laparoscopic-guided blockade, with respect to time to perform, learning curve, and postoperative analgesia. The transversus abdominis plane lies deep within the abdominal wall, potentially allowing for greater ease of access from a laparoscopic approach from within than the ultrasound guided percutaneous approach.

Prior randomized studies have been completed comparing UTAP and Placebo. In 2012 Hosgood et al. compared UTAP and placebo (UTAP w/ saline) in 46 live-donor laparoscopic nephrectomy patients (24 UTAP vs. 22 placebo). Pain control (measured using the 0-10 VAS scale) was greater on post-operative day (POD) 1 in patients receiving UTAP than in controls, 19 (15) vs. 37 (20) (presented as mean (SD)), respectively. A similar randomized study in 2014 compared UTAP and placebo (UTAP w/saline) in 21 hand assisted laparoscopic nephrectomy patients (10 UTAP vs. 11 placebo). The study was initially powered for 50 patients but with decreased accrual secondary to a surgeon taking a leave of absence during the study period. Pain scores were recorded using the 0-10 VAS score. Postoperatively at 24 hours (median (IQR)) UTAP patients demonstrated decreased postoperative pain than placebo patients (1 (0-2) vs. 4 (2-6)) on the VAS score, respectively.

A larger study, done in 2016, with 80 randomized patients undergoing retroperitoneal laparoscopic urologic surgery compared UTAP (40) and saline UTAP (40). Pain scores were assessed using the 0-100 VAS score scale. On POD1, UTAP group had lower pain scores (mean (SD)) of 8.4 (5.9) vs. placebo 28.3 (12.2).

The most recent study, done in 2018, examined 100 randomized patients undergoing robotic-assisted laparoscopic prostatectomies. Fifty patients were given UTAP blocks while the others received no block. A Numerical Rating Scale (assumed to range from 0-10 as not otherwise specified) was used to assess pain. Patients receiving the block at 24 hours had better pain control (mean (SD)) (1.8 (0.82) vs. 3.57 (0.64)).

While all of these studies point to potential efficacy of UTAP, no data has been published to date comparing laparoscopic administration of the TAP block (LTAP) to ultrasound guided administration. While these regional anesthetic blocks carry a theoretical risk of hematoma or damage to surrounding structures, none of the above studies report any complications with the injections.

The study team aims to prospectively compare Placebo (local administration), UTAP, and LTAP blocks in patients undergoing robotic surgery of the prostate and kidney. The study team expects to be able to equally efficiently administer the blocks using direct visualization and ultrasound guidance. The study team expects that a negative result would obviate the need for longer operative time by eliminating the need for the separate ultrasound guided block while a positive result would demonstrate the increased utility of preoperative ultrasound blocks in managing postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergoing Robotic Assisted Laparoscopic Partial Nephrectomy or Robotic Assisted Laparoscopic Prostatectomy
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Prior Partial Nephrectomy or Subtotal Prostatectomy Surgery (organ specific)
* Conversion to open surgery
* History of chronic pain
* History of opiate or alcohol dependence
* Allergies to local anesthetic
* Retroperitoneal surgery
* Single Port Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-02-13 (Actual); Study Completion 2021-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Mehrazin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hosgood SA, Thiyagarajan UM, Nicholson HF, Jeyapalan I, Nicholson ML. Randomized clinical trial of transversus abdominis plane block versus placebo control in live-donor nephrectomy. Transplantation. 2012 Sep 15;94(5):520-5. doi: 10.1097/TP.0b013e31825c1697. PMID 22902793
- [Background] Aniskevich S, Taner CB, Perry DK, Robards CB, Porter SB, Thomas CS, Logvinov II, Clendenen SR. Ultrasound-guided transversus abdominis plane blocks for patients undergoing laparoscopic hand-assisted nephrectomy: a randomized, placebo-controlled trial. Local Reg Anesth. 2014 May 25;7:11-6. doi: 10.2147/LRA.S61589. eCollection 2014. PMID 24860252
- [Background] Qu G, Cui XL, Liu HJ, Ji ZG, Huang YG. Ultrasound-guided Transversus Abdominis Plane Block Improves Postoperative Analgesia and Early Recovery in Patients Undergoing Retroperitoneoscopic Urologic Surgeries: A Randomized Controlled Double-blinded Trial. Chin Med Sci J. 2016 Sep 20;31(3):137-141. doi: 10.1016/s1001-9294(16)30041-4. PMID 27733219
- [Background] Dal Moro F, Aiello L, Pavarin P, Zattoni F. Ultrasound-guided transversus abdominis plane block (US-TAPb) for robot-assisted radical prostatectomy: a novel '4-point' technique-results of a prospective, randomized study. J Robot Surg. 2019 Feb;13(1):147-151. doi: 10.1007/s11701-018-0858-6. Epub 2018 Jul 28. PMID 30056612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 196 patients were eligible for the study and initially randomized. A total of 143 prostatectomy patients were deemed appropriate candidates for the trial and randomized and 114 participants were then enrolled.
  A total of 53 partial nephrectomy patients were deemed appropriate candidates for the trial. 34 participants were randomized and then enrolled.
Groups:
- Placebo/Local Anesthesia: Up to 60ml of 0.25% bupivacaine was injected directly into each of the port sites and specimen extraction site at the conclusion of the procedure prior to skin closure.
- Ultrasound-guided Transversus Abdominus Plane (UTAP) Block: 30mL of 0.25% bupivacaine administered to bilateral TAP using ultrasound guidance in prostatectomies. 40ml 0.25% aliquot bupivacaine unilateral administered in nephrectomy patients (weight based dosage permitting).
  Bupivacain: Direct injection of 0.25% bupivacaine into surgical wounds
  Ultrasound-guided transversus abdominus plane block: bilateral TAP using ultrasound guidance in prostatectomies
- Robotic -Guided Transversus Abdominus Plane (RTAP) Block: 30mL of 0.25% bupivacaine injected bilaterally in the TAP plane using a RTAP through the assistant port with a laparoscopic needle driver guidance in prostatectomies. 40ml 0.25% bupivacaine unilateral will be administered in nephrectomy patients (weight based dosage permitting).
  Bupivacain: Direct injection of 0.25% bupivacaine into surgical wounds
  Laparoscopic-guided transversus abdominus plane block: bilateral TAP using laparoscopic guidance in prostatectomies
Period: Overall Study
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Started | 28 | 64 | 56
Completed | 28 | 64 | 56
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robotic -Guided Transversus Abdominus Plane (RTAP) Block | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Placebo/Local Anesthesia | Total
Number analyzed (Participants) | 56 | 64 | 28 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.5) | 63.0 (10.6) | 63.7 (6.6) | 62.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 1 | 9
  Male | 52 | 60 | 27 | 139
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Surgical Procedure [Count of Participants; unit: Participants]
  Robotic Prostatectomy (RP) | 43 | 51 | 20 | 114
  Robotic Partial Nephrectomy (RPN) | 13 | 13 | 8 | 34
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 27.0 (4.14) | 28.6 (4.9) | 26.6 (4.25) | 27.5 (4.60)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: Visual analog scale (VAS) is a pain rating scale, with full scale from 0 to 10, higher score indicating more pain
Time Frame: 24 hours post operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Number analyzed (Participants) | 28 | 64 | 56
score on a scale | 1.29 (1.98) | 3.16 (3.10) | 2.89 (2.69)

2. Secondary Outcome: Intraoperative Time and Block Time
Description: Intraoperative time taken to complete surgical blocks and operative
Time Frame: up to 420 minutes
Measure: Median (Full Range); unit: minutes
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Number analyzed (Participants) | 28 | 64 | 56
minutes
  Time Taken to Perform Block | 2.5 [1.0 to 12.0] | 6.0 [0.5 to 14.0] | 2.5 [0.5 to 11.0]
  Total OR Time | 211.5 [137 to 293] | 224.5 [105 to 388] | 221 [114 to 419]

3. Secondary Outcome: Intraoperative Narcotic Use
Description: Intraoperative Narcotic Use in morphine equivalents
Time Frame: up to 420 minutes
Measure: Mean (Standard Deviation); unit: morphine equivalents
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Number analyzed (Participants) | 28 | 64 | 56
morphine equivalents | 27.0 (12.6) | 24.1 (12.64) | 25.5 (15.2)

4. Secondary Outcome: Intraoperative Ketoralac Use
Description: Intraoperative Ketoralac Use
Time Frame: up to 420 minutes
Measure: Median (Full Range); unit: mg
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Number analyzed (Participants) | 28 | 64 | 56
mg | 0 [0 to 30] | 0 [0 to 30] | 15 [0 to 30]

5. Secondary Outcome: Postoperative Narcotic Use
Description: Postoperative Narcotic Use in morphine equivalents
Time Frame: 24 hours post operatively
Measure: Median (Full Range); unit: morphine equivalents
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Number analyzed (Participants) | 28 | 64 | 56
morphine equivalents | 14.13 [0 to 60] | 19.50 [0 to 119] | 17 [0 to 111.50]

6. Secondary Outcome: Total Analgesic Medications
Description: The 24-hour cumulative postoperative opioid analgesic requirement was calculated using standard tables to morphine equivalents.
Time Frame: 24 hours post operatively
Measure: Median (Full Range); unit: mg morphine equivalents
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Number analyzed (Participants) | 28 | 64 | 56
mg morphine equivalents
  Acetaminophen | 1650 [650 to 5250] | 1650 [0 to 101000] | 1325 [0 to 9450]
  Ketorlac | 0 [0 to 60] | 30 [0 to 60] | 0 [0 to 90]
  Ondansetron | 0 [0 to 1] | 0 [0 to 8] | 0 [0 to 1]

7. Secondary Outcome: The Amount of Ondansetron Use
Description: Use of antiemetic medications during the postoperative course
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Number analyzed (Participants) | 28 | 64 | 56
mg | 0.05 (0.19) | 0.31 (1.30) | 0.29 (1.29)

8. Secondary Outcome: Number of Days to Return of Bowel Function
Description: Number of days to the return of bowel function
Time Frame: 2 weeks
Population: Data not collected.
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: The Length of Hospital Stay
Description: Length of hospital stay from time of surgical completion to time of discharge.
Time Frame: 2 weeks
Population: Data not collected.
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: VAS in Obese Patients
Description: 24 hour postoperative pain scores recorded using the visual analog scale (VAS) in obese patients. Visual analog scale (VAS) is a pain rating scale, with full scale from 0 to 10, higher score indicating more pain. Comparison in patients with BMI >30 and BMI<30
Time Frame: 24 hours post operatively
Population: participants divided by BMI >30 and BMI <30
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Number analyzed (Participants) | 28 | 64 | 56
score on a scale
  BMI >30: number analyzed (Participants) | 7 | 24 | 9
  BMI >30 | 1.29 (2.21) | 4.09 (2.94) | 2.33 (2.24)
  BMI <30: number analyzed (Participants) | 21 | 40 | 47
  BMI <30 | 1.29 (1.95) | 2.67 (3.11) | 3.00 (2.75)

11. Secondary Outcome: Number of Procedure Related Complications
Description: Procedure related complications and adverse events including bleeding or injection of anesthetic intravascular was determined according to Common Terminology Criteria for Adverse Events (CTCAE v 4.0).
Time Frame: 2 weeks
Measure: Number; unit: events
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
Number analyzed (Participants) | 28 | 64 | 56
events | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Placebo/Local Anesthesia | Ultrasound-guided Transversus Abdominus Plane (UTAP) Block | Robotic -Guided Transversus Abdominus Plane (RTAP) Block
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/64 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/64 | 0/56
Other Adverse Events (participants affected / at risk) | 0/28 | 0/64 | 0/56

LIMITATIONS AND CAVEATS:
This trial reflected the practice of a busy academic tertiary care center. There were numerous anesthesiologists performing the UTAP and the choice of intraoperative anesthetic and medications given was uncontrolled. In addition, multiple surgeons accrued patients to the trial with variances in operative technique. This heterogeneity among anesthesiologists and surgeons does introduce confounders but also lends to the generalizability of the present study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT04426500/Prot_SAP_000.pdf